CLINICAL TRIAL: NCT02231853
Title: Phase I/II Trial of Early Infusion of Rapidly-generated Multivirus Specific T Cells (MVST) to Prevent Post Transplant Viral Infections
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 140182; 14-H-0182
Record Dates: First submitted 2014-09-03; First posted 2014-09-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-12-29

CONDITIONS: Chronic Lymphocytic Leukemia; CML (Chronic Myelogenous Leukemia); MDS (Myelodysplastic Syndrome); Acute Lymphoblastic Leukemia; AML (Acute Myelogenous Leukemia)
Keywords: BK Virus; Cytotoxic T Cells; EBV; Adenovirus; CMV
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Adenoviridae Infections

ARMS (6):
- -1 (Experimental): 1x10e4 MVST/kg infusion
  Interventions: Biological: MVST
- 1 (Experimental): 1x10e5 MVST/kg infusion
  Interventions: Biological: MVST
- 2 (Experimental): 5x10e5 MVST/kg infusion
  Interventions: Biological: MVST
- 3 (Experimental): 1x10e6 MVST/kg infusion
  Interventions: Biological: MVST
- 3B (Experimental): 1x10e6 MVSTr/kg infusion
  Interventions: Biological: MVSTr
- 4 (Experimental): 5x10e6 MVSTr/kg infusion
  Interventions: Biological: MVSTr

INTERVENTIONS:
Biological: MVST — MVST Infusion
  Arms: -1; 1; 2; 3
Biological: MVSTr — PBMCs will be collected by apheresis prior to mobilization for Hematopoietic stem cells collection, donor apheresis will be used partially to prepare DLIs per PI specification and remaining will be further processed by elutriation.
  Monocytes and Lymphocytes are cryopreserved for further manufacture of MVSTr.
  Arms: 3B; 4

SUMMARY:
Allogeneic hematopoetic stem cell transplantation (SCT) is frequently complicated by life threatening viral reactivation. Conventional antiviral therapy is suboptimal for cytomegalovirus (CMV), adenovirus (AdV) and Epstein-Barr virus (EBV) and nonexistent for BK virus (BKV). An alternative approach to prevent viral reactivation is to infuse virus-specific cytotoxic T cells (CTL) prepared from the donor early after SCT. Such multivirus-specific CTL cells (MVST) have been successfully used in a number of centers to prevent or treat CMV, Ad and EBV. Activity of BKV-reactive cells has not been studied. Multi virus-specific T cells (MVST) are donor lymphocytes that are highly enriched for viral antigens and expanded in vitro before infusion into the transplant recipient. Viral reactivation is a particular problem inT cell depleted SCT. Median time to CMV reactivation is estimated as 28 days post T-depleted transplant, but infusion of MVST within the immediate post-SCT period has not been previously studied. This protocol will be the first of a planned series of cellular therapies to be layered on our existing T lymphocyte depleted transplant platform protocol 13-H-0144.

The aim of this study is to determine the safety and efficacy of very early infusion of MVST directed against the four most common viruses causing complications after T-depleted SCT. GMP-grade allogeneic MVST from the stem cell donor will be generated using monocyte-derived donor dendritic cells (DCs) pulsed with overlapping peptide libraries of immunodominant antigens from CMV, EBV, Ad, and BKV and expanded in IL-7 and IL-15 followed by IL-2 for 10-14 days. A fraction of the routine donor leukapheresis for lymphocytes obtained prior to stem cell mobilization will be used to generate the MVST cells. MVST passing release criteria will be cryopreserved ready for infusion post SCT.

Eligible subjects on NHLBI protocol 13-H-0144 will receive a single early infusion of MVST within 30 days (target day +14, range 0-30 days) post SCT. Phase I safety monitoring will continue for 6 weeks. Viral reactivation (CMV, EBV, Ad, BK) will be monitored by PCR by serial blood sampling. The only antiviral prophylaxis given will be acyclovir to prevent herpes simplex and varicella zoster reactivation. Subjects with rising PCR exceeding threshold for treatment, or those with clinically overt viral disease will receive conventional antiviral treatment. Patients developing acute GVHD will receive standard treatment with systemic steroids. These patients are eligible for reinfusion of MVST when steroids are tapered.

The clinical trial is designed as a single institution, open label, non-randomized Phase I/II trial of MVST in transplant recipients, designed as 3-cohort dose escalation Phase I followed by a 20 subject extension Phase II at the maximum tolerated dose of cells. Safety will be monitored continuously for a period of 6 weeks post T cell transfer. The primary safety endpoint will be the occurrence of dose limiting toxicity, defined as the occurrence of Grade IV GVHD or any other SAE that is deemed to be at least probably or definitely related to the investigational product. The primary efficacy endpoint for the phase II will be the proportion of CMV reactivation requiring treatment at day 100 post transplant. Secondary endpoints are technical feasibility of MSVT manufacture, patterns of virus reactivation by PCR, and clinical disease from EBV, Ad, BK, day 100 non-relapse mortality.

DETAILED DESCRIPTION:
Allogeneic hematopoetic stem cell transplantation (SCT) is frequently complicated by life threatening viral reactivation. Conventional antiviral therapy is suboptimal for cytomegalovirus (CMV), adenovirus (AdV) and Epstein-Barr virus (EBV) and nonexistent for BK virus (BKV). An alternative approach to prevent viral reactivation is to infuse virus-specific cytotoxic T cells (CTL) prepared from the donor early after SCT. Such multivirus-specific CTL cells (MVST) have been successfully used in a number of centers to prevent or treat CMV, Ad and EBV. Activity of BKV-reactive cells has not been studied. Multi virus-specific T cells (MVST) are donor lymphocytes that are highly enriched for viral antigens and expanded in vitro before infusion into the transplant recipient. Viral reactivation is a particular problem inT cell depleted SCT. Median time to CMV reactivation is estimated as 28 days post T-depleted transplant, but infusion of MVST within the immediate post-SCT period has not been previously studied. This protocol will be the first of a planned series of cellular therapies to be layered on our existing T lymphocyte depleted transplant platform protocol 13-H-0144.

The aim of this study is to determine the safety and efficacy of very early infusion of MVSTr cells directed against the four most common viruses causing complications after T-depleted SCT. GMP-grade allogeneic MVSTr from the stem cell donor will be generated using or peripheral blood mononuclear cells (PBMCs) pulsed with overlapping peptide libraries of immunodominant antigens from CMV, EBV, Ad, and BKV and expanded in IL-7 and IL-15 followed by IL-2 for 14 days. A fraction of the routine donor leukapheresis for lymphocytes obtained prior to stem cell mobilization will be used to generate the MVST cells. MVST passing release criteria will be cryopreserved ready for infusion post SCT.

Eligible subjects on NHLBI protocol 13-H-0144 will receive a single early infusion of MVSTr on day +7 post transplant range 0-14 days) post SCT. Phase I safety monitoring will continue for 6 weeks after infusion. Viral reactivation (CMV, EBV, Ad, BK) will be monitored by PCR by serial blood sampling. The only antiviral prophylaxis given will be acyclovir to prevent herpes simplex and varicella zoster reactivation. Subjects with rising PCR exceeding threshold for treatment, or those with clinically overt viral disease will receive conventional antiviral treatment. Patients developing acute GVHD will receive standard treatment with systemic steroids. These patients are eligible for reinfusion of MVST when steroids are tapered.

The clinical trial is designed as a single institution, open label, non-randomized Phase I trial of MVSTr in transplant recipients, designed as a single cohort Phase I study. Safety will be monitored continuously for a period of 6 weeks post MVSTr transfer. The primary safety endpoint will be the occurrence of dose limiting toxicity (DLT), defined as the occurrence of Grade IV GVHD, Grade III cytokine release syndrome (CRS), Grade III autoimmunity or any other SAE that is deemed to be at least probably or definitely related to the investigational product.

ELIGIBILITY:
* INCLUSION CRITERIA: Recipient
* Ages 18-75 years inclusive
* Patients with hematologic malignancies who have signed consent for NHLBI transplant protocol 13-H-0144.
* Susceptible to CMV reactivation post transplant (either donor or recipient need to be seropositive for CMV at any time prior to transplant).
* Ability to comprehend the investigational nature of the study and provide informed consent.

EXCLUSION CRITERIA: Recipient

* Positive pregnancy test for women of childbearing age.
* DLCO adjusted for Hb and ventilation < 50% predicted prior to SCT
* Left ventricular ejection fraction < 40% (evaluated by ECHO) or < 30% (evaluated by MUGA) prior to SCT
* AST/SGOT > 10 times ULN (>grade 3, CTCAE)
* Bilirubin > 5 times ULN (>grade 3, CTCAE)
* Estimated GFR < 15 mL/min
* Receiving Ganciclovir, Foscarnet or Cidofovir
* Receiving corticosteroids at the dose equivalent to 0.5 mg/kg/day of methylprednisolone
* Evidence of active autoimmune process

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09-03; Primary Completion 2017-11-17 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicity | 6 weeks

SECONDARY OUTCOMES:
EBV, Ad, BK, day 100 non-relapse mort. | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Minocher M Battiwalla, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gerdemann U, Keirnan JM, Katari UL, Yanagisawa R, Christin AS, Huye LE, Perna SK, Ennamuri S, Gottschalk S, Brenner MK, Heslop HE, Rooney CM, Leen AM. Rapidly generated multivirus-specific cytotoxic T lymphocytes for the prophylaxis and treatment of viral infections. Mol Ther. 2012 Aug;20(8):1622-32. doi: 10.1038/mt.2012.130. Epub 2012 Jul 17. PMID 22801446
- [Background] Walter EA, Greenberg PD, Gilbert MJ, Finch RJ, Watanabe KS, Thomas ED, Riddell SR. Reconstitution of cellular immunity against cytomegalovirus in recipients of allogeneic bone marrow by transfer of T-cell clones from the donor. N Engl J Med. 1995 Oct 19;333(16):1038-44. doi: 10.1056/NEJM199510193331603. PMID 7675046
- [Background] Blyth E, Clancy L, Simms R, Ma CK, Burgess J, Deo S, Byth K, Dubosq MC, Shaw PJ, Micklethwaite KP, Gottlieb DJ. Donor-derived CMV-specific T cells reduce the requirement for CMV-directed pharmacotherapy after allogeneic stem cell transplantation. Blood. 2013 May 2;121(18):3745-58. doi: 10.1182/blood-2012-08-448977. Epub 2013 Feb 22. PMID 23435462